CLINICAL TRIAL: NCT03845647
Title: Significance of Single Center, Open and Prospective Evaluation of Contralateral Central Lymph Node Dissection in Unilateral cN0 Differentiated Thyroid Carcinoma.
Brief Title: Significance of Contralateral Central Lymph Node Dissection in Unilateral cN0 Differentiated Thyroid Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZDWY.JRWK.002
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2019-11

CONDITIONS: Lymph Node Dissection; Lymph Node Metastases; Differentiated Thyroid Carcinoma
Keywords: lymph node dissection; differentiated thyroid carcinoma
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumor diameter<=2cm study group (Experimental): In order to provides a new theoretical basis for the operation of central lymph node in cN0 differentiated thyroid cancer,researchers are going to complete this study to evaluate the significance of contralateral central lymph node dissection in unilateral cN0 differentiated thyroid carcinoma.At the same time,it may play a certain impact on the revision of surgical guidelines for differentiated thyroid cancer.
  Interventions: Procedure: contralateral central lymph node dissection
- Tumor diameter>2cm study group (Experimental): In order to provides a new theoretical basis for the operation of central lymph node in cN0(Clinically N0) differentiated thyroid cancer,researchers are going to complete this study to evaluate the significance of contralateral central lymph node dissection in unilateral cN0 differentiated thyroid carcinoma.At the same time,it may play a certain impact on the revision of surgical guidelines for differentiated thyroid cancer.
  Interventions: Procedure: contralateral central lymph node dissection

INTERVENTIONS:
Procedure: contralateral central lymph node dissection — contralateral central lymph node dissection

SUMMARY:
There are so many contradictions over central lymph node dissection in unilateral cN0(Clinically N0) differentiated thyroid carcinoma.In order to provides a new theoretical basis for the operation of central lymph node in cN0(Clinically N0) differentiated thyroid cancer,researchers are going to complete this study to evaluate the significance of contralateral central lymph node dissection in unilateral cN0(Clinically N0) differentiated thyroid carcinoma.At the same time,it may play a certain impact on the revision of surgical guidelines for differentiated thyroid cancer.

DETAILED DESCRIPTION:
Being the most common thyroid malignant tumor,differentiated thyroid carcinoma often metastasize to the neck lymph nodes in the early stage,especially to the central lymph node.For management of cervical lymph nodes ,the 2015 American Thyroid Association Management Guidelines suggest that thyroid+Prophylactic unilateral or bilateral central lymph node dissection should be undertaken in the patients with cN0(Clinically N0) progression (T3, T4) and cN1b(Clinically N1b).Chinese guidelines recommend that, in order to avoid operative complications as far as possible (i.e. effective protection of the parathyroid gland and recurrent laryngeal nerve), lymph node dissection in the central area on the same side of the lesion should be performed at least.However, in 2017, the second edition of National Comprehensive Cancer Network(NCCN) thyroid tumor guidelines believed that if lymph nodes in the central region were negative,preventive central region lymph node dissection was not recommended.In conclusion,there are so many contradictions over central lymph node dissection in unilateral cN0 differentiated thyroid carcinoma.However,we also can draw a conclusion that it may bring some benefits if bilateral central lymph node dissection were undertaken In some cases.According to researchers' preliminary clinical trials,it is not only that there is a great probability of metastasis in the ipsilateral central lymph nodes , contralateral metastasis is also possible,and even sometimes contralateral central lymph region metastas may occur without ipsilateral central lymph nodes metastasis.In order to provides a new theoretical basis for the operation of central lymph node in cN0 differentiated thyroid cancer,researchers are going to complete this study to evaluate the significance of contralateral central lymph node dissection in unilateral cN0 differentiated thyroid carcinoma.At the same time,it may play a certain impact on the revision of surgical guidelines for differentiated thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Accurately diagnosing primary differentiated thyroid carcinoma according to pathological diagnostic criteria .

  * Differentiated thyroid carcinoma with cN0(Clinically N0) was diagnosed by thyroid ultrasound text and/or neck CT,and was confirmed with differentiated thyroid carcinoma by postoperative pathological examination.
  * The age is more than 18 years old and less than 65 years old. There is no gender restriction.
  * Untreated patients who have not received surgery, interventional therapy,chemotherapy, biotherapy, and radiation therapy.
  * Physical condition score of Eastern Cooperative Oncology Group（ECOG）: 0-2; no major organ dysfunction; oxygen partial pressure ≥ 10.64 kilopascal（kPa）; white blood cell count≥ 4 × 109/ L; hemoglobin≥ 9.5g/dL; neutrophil absolute count ≥ 1.5 × 109 / L; platelet count ≥ 100× 109 / L; total bilirubin ≤ 1.5 times of the upper limit of normal value;creatinine ≤ 1.25 times of the upper limit of normal value; and creatinine clearance ≥ 60ml / min.
  * Be able to obtain complete follow-up information, understand the situation of this study and sign informed consent.

Exclusion Criteria:

* • ①Bilateral DTC(differentiated thyroid cancer) patients ②Non-DTC(differentiated thyroid cancer)patients ③ Non-cn0(Clinically N0) patients ④ cN0(Clinically N0) patients but could not be operated on.

  * Poorly controlled diabetics (fasting blood glucose levels > 200 mg/dL). In addition to four types of malignant tumors that can be treated with radical resection, such as cervical cancer in situ, basal or squamous cell skin cancer, (breast) ductal carcinoma in situ, and organ localized prostate cancer, suffering from any other malignant tumors within 5 years.• Breastfeeding and/or pregnant women.
  * Patients with severe bleeding tendencies (prothrombin time less than 50%,cannot be corrected by treatment with vitamin K, etc.).
  * Recent severe hemoptysis, severe cough, dyspnea or patients are not able to cooperate.
  * People with severe emphysema, pulmonary congestion, and pulmonary heart disease.
  * Researchers believe that the subject may not be able to complete this study or may not be able to comply with the requirements of this study (for management reasons or other reasons).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-28 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
Tumor diameter | 12 months
  Tumor diameter will be measured by postoperative pathological examination.
Number of lymph nodes dissected in every side of central lymph node | 12 months
  Count the number of lymph nodes dissected during operation in every side of central lymph nodes of every Participants.
Number of metastatic lymph nodes diagnosed by Postoperative pathology | 12 months
  Count the number of metastatic lymph nodes diagnosed by Postoperative pathology in every side of central lymph nodes of every Participants.

SECONDARY OUTCOMES:
Rate of lymph nodes metastasis | 12 months
  Based on the statistics of Primary Outcome,count the rate of lymph node metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided